CLINICAL TRIAL: NCT05590767
Title: Department of Anesthesiology, Tri-Service General Hospital and National Defense Medical Center , Taipei, Taiwan
Brief Title: Pupillary Pain Index to Evaluate Interscalene Block and Postoperative Pain in Patients Underwent Shoulder Surgery
Status: Completed | Type: Observational
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Lu Yihsiung, Attending doctor, Department of Anesthesiology, Tri-Service General Hospital
Other Study IDs: C202205095
Record Dates: First submitted 2022-10-18; First posted 2022-10-21 (Actual); Results first posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Surgery; Shoulder Impingement
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- shoulder rotators repair: Patients scheduled to undergo shoulder rotators repair surgery
  Interventions: Procedure: Patients scheduled to undergo shoulder rotators repair surgery

INTERVENTIONS:
Procedure: Patients scheduled to undergo shoulder rotators repair surgery — Patients scheduled to undergo shoulder rotators repair surgery, and received combined general anesthesia and interscalene block

SUMMARY:
When an individual encounters nociceptive pain stimuli, the pupil dilates in a unique manner known as Pupil reflex dilation (PRD).The degree of pupillary reflex dilatation can be further quantified into an objective parameter, termed the Pupillary pain index (PPI), as a monitoring tool for the balance between nociception and antinociception in surgical patients The motivation for this study is to investigate the feasibility of using pupillometry to assess acute pain after shoulder surgery. The purpose of the study is as follows: (1) Can PDR in patients undergoing general anesthesia be used to assess the analgesic effect of interscalene block? (2) Does PPI at the end of surgical anesthesia in such patients correlate with the first numerical pain scale (NRS) during the recovery room?

DETAILED DESCRIPTION:
When an individual encounters nociceptive pain stimuli, the pupil dilates in a unique way called pupillary reflex dilation (PRD), which can be observed both when the individual is awake or under anesthesia. The degree of pupillary reflex dilatation can be further quantified into an objective parameter called the Pupillary pain index (PPI), which serves as a monitoring tool for the balance between nociception and antinociception in surgical patients. Larson studied 32 female breast surgery patients who received general anesthesia combined with thoracic paravertebral nerve block on the affected side. The results showed that the affected side of the nerve block had significantly lower pupillary reflex dilation than those without nerve block on the healthy side of the breast. The authors believed that this study confirmed the value of pupillary reflex dilation in monitoring the success rate of unilateral thoracic paravertebral nerve block during general anesthesia. In a prospective observational study of 26 patients undergoing neurosurgery under general anesthesia, Pupillary pain index at the end of surgical anesthesia and Numerical Rating Scale (NRS) during the recovery room were recorded separately, The results showed a significant correlation between the two parameters (rS = 0.62; P = 0.002). The authors concluded that the application of the measurement of pupillary reflex dilation may be useful in predicting and preventing acute postoperative pain. Shoulder rotator muscle repair is a common surgery in our hospital. Patients must receive general anesthesia, sometimes combined with scalene interscalene block (ISB), to improve postoperative acute pain ,help to perform passive shoulder rehabilitation exercises and prevent shoulder joint adhesions. Based on the above literature review, the motivation for this study was to investigate the feasibility of using pupillometry to assess acute pain after shoulder surgery. The objectives of the research project are as follows: 1. Can pupillary reflex dilation in patients undergoing general anesthesia be used to assess the analgesic effect of scalene nerve block? 2. Is the pupillary pain index (PPI) at the end of surgical anesthesia correlated with the first numerical pain scale (NRS) during the recovery room in such patients?

ELIGIBILITY:
Inclusion Criteria:

* Patients who received general anesthesia combined with ipsilateral interscalene block
* Patients listed as a Class I/II physical condition of the American Society ofAnesthesiologists

Exclusion Criteria:

* Patients younger than 20 years of age
* The presence of ophthalmologic (recent eye surgery or cataracts) or neurologic diseases (diabetic neuropathy,or postherpetic neuralgia) that could interfere with Pupillometer

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled to undergo shoulder rotators repair surgery
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-10-27 (Actual); Primary Completion 2023-08-17 (Actual); Study Completion 2023-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yeh Chun-chang, M.D., Principal Investigator — Department of Anesthesiology, Tri-Service General Hospital
Locations (1):
- Department of Anesthesiology, Tri-Service General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Shoulder Rotators Repair
Started | 40
Completed | 37
Not Completed | 3
Not completed — Protocol Violation | 1
Not completed — surgery canceled | 1
Not completed — interscalene brachial block not performed | 1

BASELINE CHARACTERISTICS:
Population: 40 patients scheduled for rotator cuff surgery were recruited for this study. Of these, three did not follow the study protocol: one had canceled surgery, one did not undergo ISB, and in one case, sevoflurane was not used as the main anesthetic. For the remaining 37 patients, Three patients did not report a loss of subjective cold/pinprick sensation in the C5 and C6 dermatomes, indicating an unsuccessful block. Therefore, 34 patients were included in the final analysis.
Arm/Group | Shoulder Rotators Repair
Number analyzed (Participants) | 34
Age, Continuous [Mean (Standard Deviation); unit: years old] | 62 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Taiwan | 34
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index (BMI) units: kg/m^2 Mean (Standard Deviation)
  kg/m^2 | 24.1 (2.7)

OUTCOME MEASURES:

1. Primary Outcome: Pupillary Pain Index (PPI )
Description: The primary outcome is the difference of the pupillary pain index (PPI ) between the ISB side and the control side The PPI mode applies a standardized, incremental transcutaneous electrical stimulation (100 Hz, 10-60mA, with 1-s intervals) that progressively increases in intensity until a pupil dilation of >13% is observed. The degree of reflex dilation is quantified on a scale of 1 (very deep analgesia) to 9 (very light analgesia) and referred to as the PPI .
Time Frame: After induction of anesthesia and before surgical incision
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Shoulder Rotators Repair
Number analyzed (Participants) | 34
score on a scale
  ISB side | 1.8 (0.2)
  Control side | 6.6 (0.3)

2. Secondary Outcome: Difference Between Intraoperative Pupillary Pain Index (PPI) and Postoperative Numerical Pain Scale (NRS)
Description: 1. PPI: The PPI mode applies a standardized, incremental transcutaneous electrical stimulation (100 Hz, 10-60mA, with 1-s intervals) that progressively increases in intensity until a pupil dilation of >13% is observed. The degree of reflex dilation is quantified on a scale of 1 (very deep analgesia) to 9 (very light analgesia) and referred to as the PPI.
  2. NRS: the nursing staff in the post-anesthesia care unit asked the patient to rate their pain at the surgical site using the NRS, with a range of 0(no pain)-10(most severe pain).
Time Frame: From emergency of anesthesia to early Post-anesthesia period
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Shoulder Rotators Repair
Number analyzed (Participants) | 34
score on a scale
  intraoperative PPI | 1.5 (0.2)
  postoperative NRS | 1.7 (1.3)

ADVERSE EVENTS:
Time Frame: 2 days
Arm/Group | Shoulder Rotators Repair
All-Cause Mortality (participants affected / at risk) | 0/34
Serious Adverse Events (participants affected / at risk) | 0/34
Other Adverse Events (participants affected / at risk) | 0/34

LIMITATIONS AND CAVEATS:
the pupillometer's built-in PPI mode utilizes electrical stimulation up to 60 mA to simulate nociception. Therefore, the patient must be under sedation or anesthesia during the measurement to ensure comfort and safety.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-20): https://cdn.clinicaltrials.gov/large-docs/67/NCT05590767/Prot_SAP_000.pdf